CLINICAL TRIAL: NCT03241823
Title: Assessment of Hepatic Fibrosis, Hemodynamics, and Disease Severity of Patients With Hepatitis C Virus Related Liver Cirrhosis After Sustained Response to Direct Acting Anti Viral Drugs.
Brief Title: Assessment of Patients With Hepatitis C Virus Related Liver Cirrhosis After Sustained Response to Direct Acting Anti Viral Drugs.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ibrahim Taha, principal investigator, Assiut University
Other Study IDs: AOHF
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Hepatitis C; Liver Cirrhosis
MeSH Terms: conditions — Hepatitis C; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hepatitis c virus related liver cirrhosis: Patients with chronic hepatitis C virus whose ultrasound shows liver cirrhosis, fibroscan "F3 and F4, Child score "A and B", of any MELD score, who achieved Sustained Virological Response after direct acting antiviral drugs (Sofosbuvir, Daclatasvir ± Ribavirin).
  Interventions: Diagnostic Test: Abdominal ultrasound .; Diagnostic Test: Model for End-Stage Liver Disease; Diagnostic Test: Fibro Scan.; Diagnostic Test: Child-Turcotte-Pugh score.

INTERVENTIONS:
Diagnostic Test: Abdominal ultrasound . — Abdominal ultrasound for each patient before and after treatment.
Diagnostic Test: Model for End-Stage Liver Disease — Model for End-Stage Liver Disease before and after treatment.
Diagnostic Test: Fibro Scan. — Liver stiffness by Fibro scan before and after treatment.
Diagnostic Test: Child-Turcotte-Pugh score. — Child-Turcotte-Pugh score before and after treatment

SUMMARY:
Hepatitis C Virus (HCV) infection is a major global health challenge; it is estimated that more than 80 million people are chronically infected worldwide, with 3-4 million new infections and 350,000 deaths occurring each year because of HCV-related complications .

DETAILED DESCRIPTION:
In 2015, a national Egyptian health issue survey was conducted to describe the prevalence of hepatitis C virus infection. The prevalence of hepatitis C virus antibody was found to be 10.0% and that of Hepatitis C virus Ribonucleic acid (HCV RNA ) to be 7.0% in the age group between 15-59 years. While In children, 1-14 years old, the prevalence of Hepatitis C virus (HCV) antibody and Hepatitis C virus Ribonucleic acid (HCV RNA) were 0.4% and 0.2% respectively.

The primary goal of HCV therapy is to cure the infection, i.e. to achieve a sustained virological response (SVR) defined as undetectable Hepatitis C virus Ribonucleic acid (HCV RNA )12 weeks or 24 weeks after treatment completion. The infection is cured in more than 99% of patients who achieve asustained virological response (SVR). Asustained virological response (SVR) is generally associated with normalization of liver enzymes and improvement or disappearance of liver necroinflammation and fibrosis in patients without cirrhosis. Patients with severe liver disease remain at risk of life-threatening complications; however hepatic fibrosis may regress and the risk of complications such as hepatic failure and portal hypertension is reduced .

Previous data suggest that the risk of Hepatocellular carcinoma and all-cause mortality is significantly reduced, but not eliminated, in cirrhotic patients who clear Hepatitis C Virus compared to untreated patients and non-sustained virological responders . Hepatitis C Virus is also associated with a number of extrahepatic manifestations and effective viral suppression induces reversal of most of them .

Studies in those with hepatitis C-related decompensated cirrhosis have demonstrated that sustained virological response can indeed be achieved in the majority of these individuals, and short-term follow-up from these studies has shown that Sustained virological response is often accompanied by improvement in measures of decompensation including Model for End-Stage Liver Disease (MELD) score and Child-Turcotte-Pugh (CPT) score. Moreover, because hepatitis C recurrence after Orthotopic liver transplantation is associated with worse outcomes, achieving Sustained virological response before transplant in a decompensated population with chronic hepatitis C will likely allow these patients to achieve long-term outcomes not different from non-Hepatitis C virus-infected populations .

In the SOLAR-1 and SOLAR-2 studies, those with decompensated cirrhosis with genotypes 1 and 4 were randomized to receive sofosbuvir/ledipasvir with low-dose ribavirin for 12 or 24 weeks . No difference was seen in Sustained virological response in the 12- or 24-week arms, and the therapy was well tolerated. Moreover, these studies both reported improvement in Model for End-Stage Liver Disease (MELD) score and Child-Turcotte-Pugh (CPT) scores 4 weeks after therapy had been stopped with longer-term follow-up results expected.

Liver stiffness measurement by transient elastography is a noninvasive, painless, rapid, and objective method for the evaluation of fibrosis or cirrhosis . Systemic reviews and meta-analyses have demonstrated the high sensitivity and specificity of Liver stiffness measurement in the diagnosis of hepatic cirrhosis.

In a systematic review conducted at 2007, repoted that at a threshold of approximately 0.60, the sensitivity and specificity of the FibroTest were 47% (35-59%) and 90% (87-92%). For FibroScan (threshold approximately 8 kPa), corresponding values were 64% (50-76%) and 87% (80-91%), respectively.

In another systematic review conducted at 2010, reported that the pooled estimates for sensitivity of fibroscan were 87% (84%-90%), specificity 91% (89%-92%) in stage IV fibrosis (cirrhosis). While in patients with stages II-IV fibrosis, they reported that the pooled estimates for sensitivity were 70% (67%-73%), specificity 84% (80%-88%).

Multicenter observational, cohort, prospective study included 90 patients with hepatitis C genotype 1 treated with telaprevir or boceprevir who had advanced fibrosis evidenced by liver stiffness and achieved Sustained virological response reported that liver stiffness was significantly reduced 2 weeks after treatment. This suggested the possibility of liver cirrhosis regression evidenced by liver stiffness after sustained virological response in a significant proportion of patients .

In a study included 182 Egyptian patients with HCV infection to validate and compare the diagnostic performance of Fibroscan , APRI Score , FIB4 for the prediction of hepatic fibrosis and treatment outcome in HCV infected patients receiving pegylated interferon and ribavirin, the authors reported that Fibroscan and noninvasive scores as APRI , FIB4 can be used as good predictors of liver fibrosis in chronic hepatitis C. However, they are not good predictors of response to pegylated interferon and ribavirin .

In a study 2010, they concluded that liver stiffness measurement can be useful for monitoring regression of liver fibrosis during entecavir treatment in patients with chronic hepatitis B virus infection.

A few studies showed a consistent relationship between Doppler Ultrasonography findings and liver histology. showed that Doppler Ultrasound findings are sensitive to haemo dynamic changes in liver fibrosis. Doppler Ultrasonography scoring was significantly related to liver fibrosis staging.

The Doppler Ultrasound signs for portal hypertension are: (1) reduced portal vein blood flow velocity (time-averaged mean vel. < 14-16 cm/s2), with sensitivity and specificity between 80-88% and 80-96%, respectively; (2) portal vein congestion index > 0.08. This parameter, however, is not used routinely, probably due to its being difficult to measure and its lower reproducibility; and (3) measurements of the hepatic arterial Resistive Index are less useful. In the course of Liver cirrhosis, the appearance of clinically significant portal hypertension worsens prognosis and Doppler ultrasound is very useful in evaluating portal hypertension. . astudy showed a significant reverse correlation between the velocities of the main portal vein and fibrous staging of the liver.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years.
2. Disease status: patients with hepatitis C Virus related liver cirrhosis child A& B (scores 5-9).
3. Previous treatment: treatment naïve and treatment experienced.
4. HCV RNA: Negative at any point between 12-24 weeks post treatment to confirm successful eradication of the virus.
5. Negative HBsAg and HIV antibody.
6. Normal kidney function test

Exclusion Criteria:

1. Child C liver cirrhosis (Child score ≥ 10).
2. HCV coinfection with HBV or HIV.
3. Patients with high risk of infection (I.V drug users, patients with blood disease requiring blood transfusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients with chronic hepatitis C virus related liver cirrhosis who achieved Sustained virological response after direct acting antiviral drugs (Sofosbuvir, Daclatasvir ± Ribavirin) and other available suitable regimens for 12 or 24 weeks will be selected from Assuit unit of treatment of viral hepatitis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Changes in liver fibrosis | 1 year.
  Using non-invasive measures "Fibroscan"

SECONDARY OUTCOMES:
Changes occurring in liver haemodynamics | 1 year.
  Using Doppler ultrasound.
Changes in severity of liver disease | 1 year
  Using Child-Pugh score.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Taha, MSc, Principal Investigator — Assiut University
Locations (1):
- Assuit Unit of Treatment of Viral Hepatitis., Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arase Y, Kobayashi M, Suzuki F, Suzuki Y, Kawamura Y, Akuta N, Kobayashi M, Sezaki H, Saito S, Hosaka T, Ikeda K, Kumada H, Kobayashi T. Effect of type 2 diabetes on risk for malignancies includes hepatocellular carcinoma in chronic hepatitis C. Hepatology. 2013 Mar;57(3):964-73. doi: 10.1002/hep.26087. Epub 2013 Feb 7. PMID 22991257
- [Background] Bruno S, Di Marco V, Iavarone M, Roffi L, Crosignani A, Calvaruso V, Aghemo A, Cabibbo G, Vigano M, Boccaccio V, Craxi A, Colombo M, Maisonneuve P. Survival of patients with HCV cirrhosis and sustained virologic response is similar to the general population. J Hepatol. 2016 Jun;64(6):1217-23. doi: 10.1016/j.jhep.2016.01.034. Epub 2016 Apr 5. PMID 27059129
- [Background] Charlton M, Everson GT, Flamm SL, Kumar P, Landis C, Brown RS Jr, Fried MW, Terrault NA, O'Leary JG, Vargas HE, Kuo A, Schiff E, Sulkowski MS, Gilroy R, Watt KD, Brown K, Kwo P, Pungpapong S, Korenblat KM, Muir AJ, Teperman L, Fontana RJ, Denning J, Arterburn S, Dvory-Sobol H, Brandt-Sarif T, Pang PS, McHutchison JG, Reddy KR, Afdhal N; SOLAR-1 Investigators. Ledipasvir and Sofosbuvir Plus Ribavirin for Treatment of HCV Infection in Patients With Advanced Liver Disease. Gastroenterology. 2015 Sep;149(3):649-59. doi: 10.1053/j.gastro.2015.05.010. Epub 2015 May 15. PMID 25985734
- [Background] Claudon M, Dietrich CF, Choi BI, Cosgrove DO, Kudo M, Nolsoe CP, Piscaglia F, Wilson SR, Barr RG, Chammas MC, Chaubal NG, Chen MH, Clevert DA, Correas JM, Ding H, Forsberg F, Fowlkes JB, Gibson RN, Goldberg BB, Lassau N, Leen EL, Mattrey RF, Moriyasu F, Solbiati L, Weskott HP, Xu HX; World Federation for Ultrasound in Medicine; European Federation of Societies for Ultrasound. Guidelines and good clinical practice recommendations for Contrast Enhanced Ultrasound (CEUS) in the liver - update 2012: A WFUMB-EFSUMB initiative in cooperation with representatives of AFSUMB, AIUM, ASUM, FLAUS and ICUS. Ultrasound Med Biol. 2013 Feb;39(2):187-210. doi: 10.1016/j.ultrasmedbio.2012.09.002. Epub 2012 Nov 5. PMID 23137926
- [Background] Enomoto M, Mori M, Ogawa T, Fujii H, Kobayashi S, Iwai S, Morikawa H, Tamori A, Sakaguchi H, Sawada A, Takeda S, Habu D, Shiomi S, Kawada N. Usefulness of transient elastography for assessment of liver fibrosis in chronic hepatitis B: Regression of liver stiffness during entecavir therapy. Hepatol Res. 2010 Sep;40(9):853-61. doi: 10.1111/j.1872-034X.2010.00687.x. PMID 20887589